CLINICAL TRIAL: NCT05351762
Title: Nimotuzumab Combined With Neoadjuvant Chemotherapy (TPF) in the Treatment of Resectable Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Nimotuzumab Combined With Neoadjuvant Chemotherapy in the Treatment of Resectable LA HNSCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPL-Nim-20210407
Record Dates: First submitted 2022-04-24; First posted 2022-04-28 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-04

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Neoadjuvant Therapy; nedaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study arm (Experimental): The study arm received nimotuzumab (400mg, every three weeks, for 2 weeks) combined with TPF chemotherapy
  Interventions: Drug: Nimotuzumab Combined With Neoadjuvant Chemotherapy

INTERVENTIONS:
Drug: Nimotuzumab Combined With Neoadjuvant Chemotherapy — The study arm received nimotuzumab (400mg, every three weeks, for 2 weeks) combined with TPF chemotherapy
  Other Names: Albumin Paclitaxel; Nedaplatin; Teggio

SUMMARY:
This study is a prospective, open-label, single-arm study. The trial will be divided into 3 phases: screening/baseline, treatment and follow-up. To initially explore the efficacy and safety of nimotuzumab combined with neoadjuvant chemotherapy (TPF regimen) in the treatment of resectable locally advanced head and neck tumors. Targeted therapy: Nimotuzumab injection 400 mg, once on the 1st day and once on the 21st day, for a total of 2 times. It should be administered by intravenous infusion 1 hour before chemotherapy, and the administration process should last for more than 60 minutes. Chemotherapy (TPF regimen): nab-paclitaxel 175mg/m2, on the 1st day; nedaplatin 100mg/m2, on the 1st day; oral administration of Sigirone on the 1st-14th day, 2/day; a treatment cycle of 21 days, a total of 2 a treatment cycle. After two cycles of chemotherapy, all patients underwent radical surgery according to whether the throat could be preserved and the patient's own wishes. The primary endpoint of the study is the tumor objective response rate (ORR), and the secondary endpoints are the primary tumor pathological complete response (pCR) rate, organ preservation rate, 1-year overall survival (OS) rate, and 1-year disease-free survival (DFS) rate. , quality of life, safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old, including 18 and 80 years old;
2. Resectable stage III to IVa head and neck squamous cell carcinoma (including oropharyngeal carcinoma, laryngeal carcinoma and hypopharyngeal carcinoma) was confirmed by histopathology or cytology by MRI imaging;
3. ECOG PS score 0-2;
4. Histopathological immunohistochemical test indicated positive EGFR expression
5. Histopathological immunohistochemical tests were P16 negative and EBER negative
6. Lymph nodes have signs of extraperitoneal invasion (MRI, CT or pathology)
7. At least one measurable lesion according to RECIST 1.1 evaluation criteria;
8. Expected survival time ≥6 months;
9. Hematologic indexes were basically normal: white blood cell count ≥4×109/L; Neutrophil absolute count ≥1.5×109/L; Platelet ≥100×109/L; Hemoglobin ≥90 g/L;
10. Normal renal function: serum creatinine ≤1.5×ULN or creatinine clearance (CrCl)> 60 mL/min(Cockcroft-Gault formula was used):

    Female CrCl=(140- age)× body weight (kg)× 0.85 / (72×Scr mg/ dL) Male CrCl=(140- age)× body weight (kg)× 1.00 / (72×Scr mg/dl)
11. Normal liver function: serum total bilirubin ≤1.5×ULN; Aspartate aminotransferase (AST) ≤2.5×ULN; Alanine aminotransferase (ALT) ≤2.5×ULN
12. Female patients must have a negative urinary pregnancy test prior to study initiation (not available in patients with bilateral oophorectomy and/or hysterectomy or postmenopausal patients)
13. Signed written informed consent.

Exclusion Criteria:

1. Received PD-1 inhibitor, EGFR mab, EGFR-TKI and anti-angiogenic drugs within 4 weeks before enrollment;
2. Participating in other interventional clinical trials within 30 days prior to screening;
3. History of other malignant tumors (except cured basal cell carcinoma of the skin)
4. there are serious and poorly controlled concurrent diseases (such as heart failure, diabetes, hypertension, liver failure, renal failure, thyroid disease, mental illness, etc.);
5. known to be infected with HIV or active viral hepatitis or tuberculosis;
6. Major surgical or planned surgery within 30 days of the first administration of the investigational drug;
7. Allergic to drugs or ingredients used in the program;
8. Women who are pregnant (as confirmed by blood or urine HCG testing) or who are lactating, or subjects of childbearing age are unwilling or unable to use effective contraceptive methods (for both male and female subjects) until at least 6 months after the last trial treatment;
9. The researcher considers it inappropriate to participate in the study;
10. Unwilling to participate in the study or unable to sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 1 year

SECONDARY OUTCOMES:
Primary pathological complete response rate (pCR) | 1 year
R0 resection rate | 1 year
Organ retention rate | 1 year
Overall survival (OS) | 1 year
Disease free survival (DFS) | 1 year
Quality of life assessed by EORTC QLQ-H&N35 | 1 year
  Quality of life assessed by EORTC QLQ-H&N35 [EORTC QLQ-H&N35 is a specific quality of life assessment scale based on EORTC QLQ-C 30, with 35 items. All of the scales and single-item measures range from 0 to 100. A high score represents a higher response level.]
Incidence of treatment-emergent adverse events | 1 year
The change of tumor related markers | 1 year
  The correlation of the value of EGFR, SCC-Ag, CEA and therapeutic effect [The changes of serum tumor markers (such as SCC-Ag and CEA were observed before and after treatment. The baseline EGFR levels on the prognosis of patients should also be explored]

IPD SHARING:
Plan to Share IPD: No